CLINICAL TRIAL: NCT07065279
Title: JY231 Injection for the Treatment of B-cell Malignancies Early Exploratory Clinical Studies on Safety, Tolerability, and Initial Efficacy
Brief Title: JY231(JY231) Injection for the Treatment of R/R B-cell Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-25-008
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: B-cell Malignancies
Keywords: B cell tumor; CAR-T; in vivo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JY231 injection for the treatment of r/r B-cell Malignancies Early exploratory clinicaltrial (Experimental): A single-center, open, single arm study JY231 Injection for the treatment of relapsed or refractory B-cell Malignancies subjects who meet the inclusion criteria will receive a single intravenous injection of JY231, followed by regular observation and follow-up of the subject.
  Interventions: Drug: JY231 Injection

INTERVENTIONS:
Drug: JY231 Injection — Patients were enrolled and given a single dose of JY231 injection intravenously, hospitalized for observation over the following month, and followed up for observation over the following 2 years.
  Other Names: in vivo CAR-T

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with relapsed or refractory B-cell Malignancies.

It is an early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of relapsed or refractory B-cell Malignancies.

DETAILED DESCRIPTION:
This is an open-label, single-arm study to evaluate the efficacy and safety of in vivo Chimeric Antigen Receptor T-Cell(CAR-T cell) therapy in patients with relapsed refractory B-cell Malignancies. Upon enrollment, subjects will receive an intravenous infusion of the JY231 preparation. Following the infusion, subjects will be hospitalized for one month for observation, and subjects will be evaluated for safety and efficacy. Subjects will be followed for up to 2 years to determine if the disease is under control.

ELIGIBILITY:
Inclusion Criteria:

1. up to 75 years (Child, Adult) , either sex, sign informed consent (ICE);
2. Histologically confirmed as B-cell Malignancies ;
3. Flow cytometry or histology confirmed positive expression of cluster of differentiation 19(CD19);
4. According to the researcher's assessment, the expected survival period is greater than 3 months;
5. Eastern Cooperative Oncology Group(ECOG) physical condition score ≤ 3;
6. The patient has good liver, kidney, heart, and lung functions: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal(ULN), which can be relaxed to ≤ 5 × ULN for patients with liver invasion; Total serum bilirubin # 34 μ Mol/L; Creatinine clearance rate>30 mL/min; Cardiac ejection fraction (EF) ≥ 40%, without pericardial effusion and significant arrhythmia; Indoor oxygen saturation(SpO2) ≥ 92%;
7. Peripheral blood lymphocyte absolute count: absolute lymphocyte count(ALC) ≥ 0.5 × 109/L, blood platelet(PLT)>30 × 109/L, Hb>80 g/L, with a single venous access and no other contraindications for blood cell separation;
8. Individuals with fertility must agree to the use of efficient contraceptive methods;
9. The subject or their legal guardian can understand and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women, as well as women with pregnancy plans within six months;
2. Virological tests of hepatitis B, hepatitis C, AIDS, syphilis and cytomegalovirus were positive;
3. Having a history of other tumors (excluding skin or cervical carcinoma in situ cured by root therapy and without evidence of disease activity);
4. Previously received treatment targeting CD19;
5. Received autologous hematopoietic stem cell transplantation within 6 weeks;
6. The presence of uncontrollable active bacterial or fungal infections;
7. Allergies to research related drugs or cellular components;
8. Active autoimmune diseases exist;
9. Patients with unstable or active ulcers or gastrointestinal bleeding currently present;
10. Individuals with mental or psychological disorders who cannot cooperate with treatment and efficacy evaluation;
11. Received other experimental drug treatments within the past 3 months;
12. Existence of grade II-IV acute graft versus-host disease(GVHD) or widespread chronic GVHD;
13. Researchers believe that other reasons are not suitable for clinical trial participants.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.
Incidence of adverse events(AE) after infusion | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.

SECONDARY OUTCOMES:
Objective Response Rate | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  Objective Response Rate(ORR) is defined as the proportion of subjects achieving complete remission(CR) and partial response(PR).

CONTACTS AND LOCATIONS:
Locations (1):
- 920th HJointLogistics, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No